CLINICAL TRIAL: NCT05940818
Title: The Effect Thirsty and Oral Care Frequency of Cold Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, SERAP GÜNGÖR, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Thisrty
Record Dates: First submitted 2023-07-02; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Thirst
Keywords: Postoperative Period; ice; nursing; thirst; Intensive care units; mouth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): In the study group, the intensive care oral care frequency assessment scale was applied to 55 patients at the end of the 16th hour, in addition to the assessment of pain and thirst at the 1st, 4th, 8th, and 16th hours postoperatively. In patients with a thirst of 3 and above, the bedside was lifted 30-450 times (to prevent bronchoaspiration), and cold water spray (kept in the refrigerator at +4°C and stored) was sprayed 3 times (approximately 2 ml) into the mouth of the patient every hour. Evidence suggests that the risk of bronchoaspiration is minimal up to the 50 mL and 1.5 mL/kg limit of gastric volume (Doi et al., 2021). For this, it is thought that the application of an average of 32 ml of cold water applied to the patients is reliable. The standard oral care of the clinic was applied to the patients who needed oral care. It was also recorded how many times oral care was given to the patients included in the study within 16 hours.
  Interventions: Behavioral: the intensive oral care
- control group (No Intervention): In the control group, standard nursing care was applied to 55 patients with the pain, thirst and intensive care oral care frequency assessment scale at the 1st, 4th, 8th, and 16th hours postoperatively.

INTERVENTIONS:
Behavioral: the intensive oral care — the intensive oral care
  Arms: experimental group

SUMMARY:
Surgical patients, and especially bariatric patients, are high-risk patients who may develop thirst due to intubation, blood loss, osmotic imbalance, and prolonged fasting. Nurses often have the perception that when the patient's oral intake is turned off, nothing can be done to prevent thirst and dry mouth. Thirst is one of the main stress factors that reduces the comfort of intensive care patients. So far, no assessment has been routinely used to assess thirst and dry mouth. However, thirst is a mitigable symptom that should be evaluated by the nurse.

DETAILED DESCRIPTION:
The data were collected by the researcher by face-to-face interview technique between April 2022 and March 2023 in the groups participating in the study. It was applied to patients who agreed to participate by giving information about the purpose of the study to patients who met the research criteria. The patients were divided into 2 groups as study and control. In the study group, the intensive care oral care frequency assessment scale was applied to 55 patients at the end of the 16th hour, in addition to the assessment of pain and thirst at the 1st, 4th, 8th, and 16th hours postoperatively. It was applied to patients with a thirst of 3 and above by spraying cold water into the mouth of the patient every hour. The standard oral care of the clinic was applied to the patients who needed oral care. In the control group, standard nursing care was applied to 55 patients with the pain, thirst and intensive care oral care frequency assessment scale at the 1st, 4th, 8th, and 16th hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18-65, Level of consciousness (level A of AVPU) and orientation (place, direction, time) swallowing and coughing reflex without nausea-vomiting No mandible fracture No dialysis treatment When we ask about their thirst, those who have 3 or more thirst on a scale of 0-10 hungry for more than 6 hours Anesthesia duration exceeding 1 hour Patients not receiving Mechanical Ventilator support undergoing elective surgery Individuals who can communicate at a level that can answer the research questions will be included.

Those who do not use dentures

Exclusion Criteria:

* be over 65, under 18 Having lesions on the oral mucosa and lips Having any disease that prevents communication such as Alzheimer's, dementia Patients with a thirst feeling of 3 or less during the cold spray application

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 55 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Study Group Outcome | 16 hours
  In the study group, 55 patients were evaluated for pain and thirst at the 1st, 4th, 8th and 16th postoperative hours and the intensive care oral care frequency assessment scale was additionally applied at the end of the 16th hour without oral care.
Control Group Outcome | 16 hours
  In the control group, standard nursing care was applied to 55 patients at the 1st, 4th, 8th, 16th postoperative hours with the intensive care oral care frequency assessment scale at the end of the 16th hour without pain, thirst and oral care.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No